CLINICAL TRIAL: NCT04676230
Title: Effectiveness of an ICCMS™ Caries Management Program. A Schoolchildren Multicenter Randomized Controlled Trial.
Brief Title: Effectiveness of an ICCMS™ Caries Management Program.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad El Bosque, Bogotá (Other)
Responsible Party: Principal Investigator, Stefania Martignon, Principal Investigator, Universidad El Bosque, Bogotá
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 008-2014
Record Dates: First submitted 2019-05-10; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Caries
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): caries management based on the ICCMSTM: Patient intervention according to the caries risk likelihood: high, moderate or low. Surfaces intervention according to the surface diagnosis decision matrix (ICCMSTM): Mi: Initial caries management, Mm: Moderate caries management, and Me: Extensive caries management.
  Interventions: Procedure: Experimental group
- Control group (Active Comparator): Systematic patient caries risk intervention (all managed as high risk patients). Surfaces intervention with conventional caries management of cavitated/dentin caries lesions (restorative treatment).
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Experimental group — Caries management based on the ICCMSTM: Patient intervention according to the caries risk likelihood: high, moderate or low. Surfaces intervention according to the surface diagnosis decision matrix (ICCMSTM): Mi: Initial caries management, Mm: Moderate caries management, and Me: Extensive caries management.
  Other Names: ICCMS™ group
  Arms: Experimental group
Procedure: Control group — Systematic patient caries risk intervention (all managed as high risk patients). Surfaces intervention with conventional caries management of cavitated/dentin caries lesions (restorative treatment).
  Other Names: Colombian Health System
  Arms: Control group

SUMMARY:
The aim of this study is to compare in schoolchildren the effectiveness of an updated caries management program based on the current caries paradigm with the ICCMS™ system (International Caries Classification and Management System) versus an adjusted Colombian dental public health service caries management program, in terms of: 1- caries risk probability, 2- caries lesions, 3- parents' knowledge, attitudes and practices regarding children's oral health.

Null hypothesis: the caries management program based on its current paradigm offers the same degree of effectiveness than the conventional caries management program.

Alternative hypothesis: the caries management program based on its current paradigm offers a different degree of effectiveness than the conventional caries management program.

DETAILED DESCRIPTION:
This study counts with ethical approval from the Ethics Board in Universidad El Bosque (UEB 008-2014).

Population:

The study population will be 6-7 year-old schoolchildren from the six participant dental schools.

Baseline examination:

The baseline examination will be conducted by the site coordinator examiner. Once the informed consent is signed by the parents and the children give their acceptance, a comprehensive examination will be performed, including:

* Parents' knowledge, attitudes and practices survey regarding children's oral health.
* Caries risk probability assessment through individual caries risk assessment plus patient current caries status: low, moderate, high.
* Radiographic caries detection using the ICCMS™ criteria.
* Clinical examination:

  * dmf/DMF T/S
  * PUFA Index
  * Dental surface restoration conditions
  * ICCMS™ caries visual detection: Cs: Sound Surfaces (ICDAS code 0); Ci: Initial-stage caries lesion (ICDAS codes 1 y 2); Cm3/Cm4: Moderate-stage caries lesion (ICDAS codes 3-microcavity y 4-dentin shadow) and Ce: Extensive-stage caries lesion (ICDAS codes 5 y 6)
* Progression assessment of present caries lesions using ICCMS™ criteria in terms of Active or Inactive.

Synthesis and analysis:

The synthesis and analysis of the gathered information will conduce to the ICCMS™ caries management decision plan in terms of caries risk likelihood management and caries lesions management with a structure conservative approach.

This study counts with ethical approval from the Ethics Board in Universidad El Bosque (UEB 008-2014).

Population:

The study population will be 6-7 year-old schoolchildren from the six participant dental schools.

Baseline examination:

The baseline examination will be conducted by the site coordinator examiner. Once the informed consent is signed by the parents and the children give their acceptance, a comprehensive examination will be performed, including:

* Parents' knowledge, attitudes and practices survey regarding children's oral health.
* Caries risk probability assessment through individual caries risk assessment plus patient current caries status: low, moderate, high.
* Radiographic caries detection using the ICCMS™ criteria.
* Clinical examination:

  * dmf/DMF T/S
  * PUFA Index
  * Dental surface restoration conditions
  * ICCMS™ caries visual detection: Cs: Sound Surfaces (ICDAS code 0); Ci: Initial-stage caries lesion (ICDAS codes 1 y 2); Cm3/Cm4: Moderate-stage caries lesion (ICDAS codes 3-microcavity y 4-dentin shadow) and Ce: Extensive-stage caries lesion (ICDAS codes 5 y 6)
* Progression assessment of present caries lesions using ICCMS™ criteria in terms of Active or Inactive.

Synthesis and analysis:

The synthesis and analysis of the gathered information will conduce to the ICCMS™ caries management decision plan in terms of caries risk likelihood management and caries lesions management with a structure conservative approach.

The first step of the management plan considers the caries risk likelihood.

The management options include:

* Low likelihood: Tooth brushing 2/day with a fluoride toothpaste (≥1,000 ppm F-), following the dental team instructions; motivational engagement (discuss with patients how to improve oral health behaviors - including amount of sugar); cross-brushing for erupting first molars; use of dental floss; recalls every 6 months, including professional cleaning.
* Moderate likelihood: Previous activities plus prescribed F- mouthrinse; sealants in caries risk surfaces, F- varnish 2 times/year; motivational interviewing; recalls every 3 months, including professional cleaning.
* High likelihood: Previous activities and increase F- varnish to 4 times/year plus Topical F- application; counseling: reduce sugar amount & frequency; recalls every 3 months, including professional cleaning.

The patient's caries risk factors management plan is tailored at the individual level and involves actions to protect sound tooth surfaces from developing new caries lesions, and all current active and inactive lesions from progressing. In addition, it aims at lowering the caries risk likelihood of the patient when moderate or high, and to maintain it if low.

The second step is the caries diagnosis decision making at the surface level which conducts to the surface diagnosis decision matrix. This decision relies on the clinical classification of dental caries using ICCMS™ criteria and the radiographic extent of the lesion (enamel or dentin) plus the activity status of the lesions. Only active caries lesions require caries management. The level of intervention depends on the clinical caries classification of the surface or tooth and the radiological extent (when information is available) of the lesion in enamel or dentin. Management levels of active caries lesions are classified as follows:

* MInitial: Initial caries management stage (non-operative care (NOC)-control)
* MModerate: Moderate caries management stage (minimally invasive surgical caries management with no or minimal dentin removal)
* MExtensive: Extensive caries management stage (invasive surgical caries management with dentin removal).

For sound surfaces, risk based prevention is performed. For inactive lesions, restorations might be performed depending on esthetic and plaque retention reasons.

Intervention:

The children will be randomized in two groups as follows:

Group A (Experimental): ICCMS™ caries management according to the surface diagnosis decision matrix of active Ci, Cm3/4, and Ce caries lesions. Individual management according to the future patient caries risk likelihood with specific prevention strategies.

Group B (Control): conventional caries management. Operative treatment of Cm and Ce caries lesions (caries shadows and cavities) with conventional restorative treatment. Systematic caries risk management with twice-a-year fluoride gel application, sealants on all occlusal surfaces and oral health literacy.

When the management plan is finalized in both groups, patients must continue attending the clinic according to their group for the following three years.

Follow-up assessments will be conducted at one and three years after baseline, with the baseline indicators as described above.

ELIGIBILITY:
Inclusion Criteria:

* Children from 6 to 7 years old
* Informed consent signed
* Children in standard good general health

Exclusion Criteria:

* Children with physical disability and/or cognitive diseases
* Children whose family will is planning to move from the city in the following 36 months
* Children with orthopedic/orthodontic appliances at baseline

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Evolution of ICCMSTM caries likelihood after 1 and 3 years. | up to 36 months
  Change in ICCMSTM caries likelihood subjects' distribution after 1 and 3 years

SECONDARY OUTCOMES:
Presence of new caries lesions in terms of ICCMSTM categories after 1 and 3 years. | up to 36 months
  Change in the presence of new caries lesions in terms of ICCMSTM categories after 1 and 3 years.
Number of appointments after 1 and 3 years. | up to 36 months
  Total number of appointments after1 and 3 years.
Progression of existing caries lesion in terms of ICCMSTM categories after 1 and 3 years. | up to 36 months
  Change in the progression of existing caries lesion in terms of ICCMSTM categories after 1 and 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Martignon, PhD, Principal Investigator — UNICA - Unidad de Investigación en Caries, Facultad de Odontología
Locations (1):
- Universidad El Bosque, Bogotá, D.C:, Colombia